CLINICAL TRIAL: NCT06071091
Title: Comparison of Permanent Intracranial Stenting Versus no Stenting in Stroke Secondary to Refractory Acute Proximal Vascular Occlusion: a Multicenter Randomized Controlled Trial
Brief Title: Permanent Intracranial Stenting for Acute Ischemic Stroke Related to a Refractory Large Vessel Occlusion
Acronym: PISTAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP210091; 2022-A00570-43 (Other: ID-RCB)
Record Dates: First submitted 2023-09-04; First posted 2023-10-06 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Brain; Intracranial; Ischemia; Stroke; Mechanical Thrombectomy; Intracranial Occlusion; Refractory Occlusion; Interventional; Angioplasty; Stenting
MeSH Terms: conditions — Ischemic Stroke; Ischemia; Stroke; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracranial stenting (Experimental): Rescue Intracranial Stenting + best medical treatment
  Interventions: Device: Intracranial stenting
- Best medical management alone (Active Comparator): Best medical treatment with no additional thrombectomy passes
  Interventions: Other: Optimal medical care, without additional endovascular procedures

INTERVENTIONS:
Device: Intracranial stenting — In order to promote the efficacy of the stent to reopen the target vessel, there are two requirments prior stenting: First, balloon angioplasty can be performed at operators' discretion based on angiographic findings. Second, a dual antiplatelet therapy protocol is considered essential to maintain stent patency, and therefore should be introduced before stent implantation whenever possible.
  Permanent Intracranial can then be performed according to the standard technique: An autoexpandable intracranial stent (Neuroform Atlas 4x24mm) is deployed though a dedicated microcatheter over the target refractory occlusion The only stent system allowed is the Neuroform Atlas 4x24mm (Stryker Neurovascular) The anti-thrombotic drugs used, their route of administration, the choice of navigation equipment are left to the discretion of the team in charge of the patient. A standardized anti-thrombotic protocol will be proposed as an indication.
  Arms: Intracranial stenting
Other: Optimal medical care, without additional endovascular procedures — The control group represents the standard therapeutic strategy for refractory vascular occlusions, which consists of stopping the procedure without performing any additional mechanical thrombectomy attempts.
  In this group, the procedure will be stopped after randomization and a control seriography will be performed to confirm the persistent nature of the intracranial occlusion.
  The patient will benefit from the best medical care available, which may include any medical treatment including a dual anti-platelet therapy if the therapeutic team deems it necessary (Standard medical care may also include (non-exhaustive list):
  * Nursing
  * Nursing care
  * Symptomatic treatments: analgesics for example
  * Systematic clinical monitoring and control imaging if necessary
  * Rehabilitation if necessary)
  Arms: Best medical management alone

SUMMARY:
Clot extraction failure during mechanical thrombectomy is a major concern in the management of acute ischemic stroke related to large vessel occlusions. Indeed, it can occur in up to 10 to 30% of cases and, therefore, is associated with a very poor prognosis. These refractory occlusions frequently occur when an underlying intracranial atherosclerotic disease is present. Thus, one of the most promising rescue technique consists of placing a permanent intracranial stent, under dual antiplatelet therapy over the target refractory occlusion. This strategy is well studied in coronary occlusions where the atheroscotic mechanism is highly prevalent. However, as the ischemiated brain is at much higher risk of hemorrhagic complications, such strategy entails a greater risk. This raises the question of whether such risk is worth the reward of obtaining reperfusion. The investigators designed this randomized study in order to evaluate whether a strategy combining rescue pemanent intracranial stenting with the best medical treatment is superior to the best medical treatment alone in acute refractory large vessel occlusions.

DETAILED DESCRIPTION:
These past recent years, mechanichal thrombectomy has become the standard treatment for acute ischemic strokes due to large vessel occlusions. Mechanical thrombectomy failure occurs in about 10 to 30% of cases with disastrous consequences for these patients. Indeed, reperfusion failures are associated with 30.5% mortality rates and only 21% of all patients are able to achieve functional independence at 3 months.

In order to treat these refractory large vessel occlusions many techniques and devices have been developped. Rescue Intracranial Stenting (RIS) is the most studied technique and the most promising one. However, RIS requires strong antithrombotic medications to ensure stent patency, which may increase the risk of hemorrhagic complications.

The investigators recently performed a meta-analysis of observational data, that showed that RIS in refractory large vessel occlusions allowed significant improvements in functional outcome at 3 months. The rate of good functional outcome at 3 months went from 21% in the control group (no RIS) to 43% in the RIS group. Mortality was also significantly reduced from 30.5% (control group) to 18.8% in the RIS group. Furthermore, RIS did not increase the rate of symptomatic intracranial hemorrhage.

Of course, this meta-analysis is only based on observational data and needs to be confirmed in a randomized trial to bring the highest level of evidence.

Refractory large vessel occlusions are commonly caused by an underlying intracranial atherosclerotic plaque. Since the SAMMPRIS trial, most of the indications for the endovascular treatment of intracranial atherosclerotic stenoses have been removed. Nevertheless, there are subsets of patients who actually benefit from intracranial stenting such as patients with refractory large vessel occlusions or patients with hemodynamically significant stenoses. As such, the PISTAR trial could be a way of validating intracranial stenting in this indication.

All patients admitted for a mechanical thrombectomy will be screened before the procedure. If the patient fulfills the preoperative elligibility criteria, she/he will be informed of the possibility of being included in case of a refractory occlusion. If the patients' clinical state does not allow her/him to give informed consent, she/he can still be included using an emergency consent procedure. Consents to pursue the study will be sought as soon as possible, from the patient or her/his trusted relative.

If the patient meets all remaining elligibility criteria during the mechanical thrombectomy in particular if the occlusion is considered as refractory, she/he can be included and randomized.

Randomization will be performed using a minimization procedure based on the recruiting center, the administration of IV thrombolysis and the location of the occlusion (anterior versus posterior circulation). The randomzation will be centralized using an online e-crf platform.

The patient can be randomized in one of the two following arms

* Intervention arm : RIS + best medical treatment In this arm, a dedicated antithrombotic protocol will be initiated before the deployment of the stent. The choice of antithrombotics and the need to perform additional endovascular manœuvres such as balloon angioplasty will be left at the operator's discretion. A standard protocol for antithrombotics is proposed.
* Control arm : best medical treatment with no additional thrombectomy passes In this arm, the procedure is stopped and a last control angiogram is performed to confirm the absence of reperfusion. Any additional medical treatment is allowed.

Follow up visits will be performed immediately after the procedure (V0), at 24hrs (V1), 72hs (V2) and 1 month (V3). The end-research visit will be performed at 3 months (+/- 15 days) and a remote safety visit will be performed at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Acute ischemic stroke secondary to an occlusion of the internal carotid artery termination OR the 1st or 2nd segment of the middle cerebral artery OR the basilar artery and/or the 4th segment of the vertebral artery radiologically proven (CT Angiography or angio-MRI)
* Patient within the authorised timeframe for a MT, according to the AHA/ASA 2019 grade I recommendations
* Refractory intracranial large vessel occlusion defined as :

Persistent arterial occlusion (mTICI 0 or I) after a minimum of 3 mechanical thrombectomy passes using direct aspiration or a stent retriever OR Early arterial reocclusion (<10 minutes) after at least one pass OR Underlying stenosis (estimated between 70 and 99%)

* ASPECT Score for CT or DWI-ASPECTS for MRI or pc(-DWI)- ASPECTS (posterior circulation) ≥ 5
* Independent patient before stroke (mRS 0-2)
* Patient's or her/his trusted relative's consent or emergency procedure consent

Exclusion Criteria:

* Proximal intracranial vascular occlusion not confirmed on angiography
* Intracranial bleeding <3 months or intracranial bleeding during TM procedure prior to inclusion
* Contraindication to a dual antiplatelet therapy
* Mechanical thrombectomy procedure requiring carotid or vertebral arterial access by direct puncture
* Proof of significant ischemic lesions in a vascular territory not affected by the occlusion
* Proven allergy to iodinated contrast material
* Patient known for severe renal impairment with creatinine clearance < 30ml/min
* Pregnant or breastfeeding women
* Tandem occlusion (defined as the association of an intracranial occlusion to a cervical steno-occlusive lesion on the same arterial axis that needs additional endovascular manœuvers for the cervical lesion)
* Major comorbidities that could hinder the improvement or the follow up of the patient or the benefit of the intervention
* Unaffiliation to the French Social Security system
* Patient under juridic protection
* Patient participating in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of independent patients | 3 months
  Rate of independent patients at 3 months, defined as a modified Rankin Scale (mRS) 0-2, evaluated by a trained health professional, blinded to the randomization arm.
  Min=0 ; Max=6 (lower is better)

SECONDARY OUTCOMES:
Mortality | 6 months
  Mortality rate at 6 months
Excellent functional outcome | 3 months
  Rate of excellent functional prognosis defined as a modified Rankin Scale (mRS) score of 0-1 at 3 months Min=0 ; Max=6 (lower is better)
modified Rankin Scale (mRS) | 3 months
  Distribution of mRS scores at 3 months Min=0 ; Max=6 (lower is better)
Successful reperfusion | End of procedure (up to 4 hours)
  Successful reperfusion rate (Score modified Thrombolysis In Cerebral Infarction [mTICI] ≥IIb) Min=0 ; Max=3 (higher is better)
Excellent reperfusion | End of procedure (up to 4 hours)
  Excellent reperfusion rate (defined as modified Thrombolysis In Cerebral Infarction [mTICI] score ≥IIc) Min=0 ; Max=3 (higher is better)
Symptomatic ischemic recurrence | 3 months
  Rate of symptomatic ischemic recurrence (≥4 points of National Institutes of Health Stroke Scale (NIHSS) compared to the lowest NIHSS score during management) certified by imaging within 3 months.
  Min=0 ; Max=42 (lower is better)
Rate of patients requiring a new mechanical thrombectomy | 3 months
  Rate of patients requiring a new mechanical thrombectomy within the group of patients with symtomatic ischemic recurrence
Neurologic recovery | 24 hours
  Neurologic recovery at 24 hours, according to the National Institutes of Health Stroke Scale (NIHSS) score as compared to initial NIHSS score Min=0 ; Max=42 (lower is better)
Neurologic recovery | 72 hours
  Neurologic recovery at 72 hours, according to the National Institutes of Health Stroke Scale (NIHSS) score as compared to initial NIHSS score Min=0 ; Max=42 (lower is better)
Periprocedural time (time between arterial puncture and successful reperfusion (if obtained)) | End of procedure (up to 4 hours)
  Time between arterial puncture and successful reperfusion (if obtained)
Periprocedural time (Time between onset of symptoms (or "last seen normal") and successful reperfusion (if obtained)) | End of procedure (up to 4 hours)
  Time between onset of symptoms (or "last seen normal") and successful reperfusion (if obtained)
Periprocedural time (Time between randomization and successful reperfusion (if obtained)) | End of procedure (up to 4 hours)
  Time between randomization and successful reperfusion (if obtained)
Procedure duration | End of procedure (up to 4 hours)
  Time between arterial puncture and arterial closure
Intracranial hemorrhagic complications | 6 months
  Rate of symptomatic intracranial haemorrhage at 6 months defined as any intracranial haemorrhage responsible for neurological deterioration (≥4 NIHSS points compared to the lowest NIHSS score during management)
Distribution of intracranial hemorrhagic complications | 6 months
  Distribution of intracranial hemorrhagic complications according to the Heidelberg classification
Serious extracranial hemorrhagic complications | 6 months
  Rate of serious extra-cranial hemorrhagic complications at 6 months, defined as any extra-cranial bleeding complication requiring re-hospitalization and/or surgery and/or blood transfusion
All procedural complications | Up to 6 months
  Rate of all procedural complications, including vascular perforation, dissection, embolism in a territory not previously affected by the ischemia and serious complications on the arterial access (as defined below)
Vascular perforation | End of procedure (up to 4 hours)
  Rate of vascular perforation during the procedure
Dissection | End of procedure (up to 4 hours)
  Rate of dissection during the procedure
Embolism in a territory not previously affected by the ischemia | End of procedure (up to 4 hours)
  Rate of embolism in a territory not previously affected by the ischemia, during the procedure
Serious complication on the arterial access | 6 months
  Rate of serious complications on the arterial access, defined as any superficial hematoma with deglobulisation [loss of 2 Hb points on the NFS] and/or requiring a transfusion, retroperitoneal hematoma with or without deglobulisation, arterial pseudo-aneurysm at the puncture site requiring surgical treatment, femoral artery occlusion and/or acute limb ischemia, puncture site abscess.
Vascular reocclusion | 24 hours
  Rate of vascular reocclusion on 24-hour imaging
Adverse events | 6 months
  Rate of adverse events at 6 months
Serious adverse events | 6 months
  Rate of serious adverse events at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin PREMAT, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (12):
- France (12):
  - CHU Amiens, Amiens
  - CHU Bordeaux (Pellegrin Hospital), Bordeaux
  - Henri-Mondor Hospital (APHP), Créteil
  - Bicêtre Hospital (AP-HP), Le Kremlin-Bicêtre
  - Bicêtre Hospital (APHP), Le Kremlin-Bicêtre
  - CHU Lille (Roger Salengro Hospital), Lille
  - CHU Montpellier - Gui de Chauliac, Montpellier
  - CHRU de Nancy, Nancy
  - Lariboisière Hospital (APHP), Paris
  - APHP • Assistance Publique des Hôpitaux de Paris, Pitié-Salpêtrière hospital, Paris
  - CHU Poitiers, Poitiers
  - Foch Hospital, Suresnes

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Premat K, Dechartres A, Baptiste A, Guedon A, Mazighi M, Spelle L, Denier C, Tuilier T, Hosseini H, Lapergue B, Di Maria F, Bricout N, Henon H, Gory B, Richard S, Chivot C, Courselle A, Velasco S, Lamy M, Costalat V, Arquizan C, Marnat G, Sibon I, Lenck S, Shotar E, Allard J, Sourour N, Degos V, Alamowitch S, Clarencon F. Comparison of rescue intracranial stenting versus best medical treatment alone in acute refractory large vessel occlusion: study protocol for the PISTAR multicenter randomized trial. J Neurointerv Surg. 2025 Mar 17;17(4):360-367. doi: 10.1136/jnis-2024-021502. PMID 38538057